CLINICAL TRIAL: NCT04123925
Title: Preoperative Nivolumab in Patients With Locally Advanced Colon Cancer (T3 or T4): a Window-of-opportunity Study
Acronym: NICOLE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NICOLE
Record Dates: First submitted 2019-09-04; First posted 2019-10-11 (Actual); Last update posted 2020-06-12 (Actual); Status verified 2019-09

CONDITIONS: Colon Cancer Stage II/III
Keywords: locally advanced colon; neoadjuvant; nivolumab
MeSH Terms: interventions — Nivolumab; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nivolumab (Experimental): Patients will receive nivolumab at a flat dosage of 240 mg every two weeks on Day -28 and Day-14 (+/- one day) prior to planned surgery on Day 0 or up to +7 days
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab — Locally advanced colon cancer must be documented at screening (within 21 days prior to initiation of study treatment) and re-assessed prior surgery by spiral or multidetector computed tomography (CT) scan Postoperatively, standard adjuvant chemotherapy will be administered in pathological III-stage and at investigator discretion in pathological II-stage at high risk
  Other Names: Surgery

SUMMARY:
A monocentric window of opportunity study preceded by a safety run-in phase. The study population will include locally advanced colon patients (T3 or T4).

DETAILED DESCRIPTION:
An initial 6-patients safety run-in cohort will be followed by an expansion cohort, with a planned accrual of 16 patients.

Patients will receive nivolumab at a flat dosage of 240 mg every two weeks on Day -28 and Day-14 (+/- one day) prior to planned surgery on Day 0 or up to +7 days. Locally advanced colon cancer must be documented at screening (within 21 days prior to initiation of study treatment) and re-assessed prior surgery by spiral or multidetector computed tomography (CT) scan.

Postoperatively, standard adjuvant chemotherapy will be administered in pathological III-stage and at investigator discretion in pathological II-stage.

Safety Assessments: Toxicities will be evaluated throughout the study treatment and up to 30 days after surgery. Toxicity will be graded according to the NCI Common Toxicity Criteria.

The National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI CTC-AE) Version 4.03 will be used to evaluate the clinical safety of the treatment in this study. Patients will be assessed for AEs at each clinical visit and as necessary throughout the study. Grade ≥3 hematological and non-hematological toxicities will be recorded.

Efficacy Assessments: Pathological tumor regression will be evaluated according to Mandard modified scoring system [Mandard 1994].

Biomarker study: The Immunoscore evaluation will be assessed using standardized Immunoscore assays and software (HalioDx).

Additional correlative biological studies will be performed for the evaluation of the biomarkers indicated above on the biological samples (paraffin-embedded tissue, frozen tissue, blood, serum, etc.). Biomarkers will be evaluated on tumor tissues obtained by biopsies at baseline, and by surgery after neoadjuvant treatment. A comparison with a subsequent cohort of 22 patients with locally advanced colon cancer (T3-T4) who proceed to surgical resection without preoperative anti-PD-1 and recruited following the end of the enrollemnt of the planned pateints in the Nicole study, will be performed.

Blood samples will be collected at baseline, prior to surgery, and at the recurrence of the disease (progressive disease [PD]). Biomarkers will be correlated with pathological response and patient's outcome.

Patients will have follow-up evaluation every six months for five years.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with histologically confirmed adenocarcinoma of colon with staging of locally advanced (T3 or T4)
2. No prior treatments (chemotherapy, radiation or surgery) for colon cancer
3. Either sex aged ≥ 18 years
4. Colon lesion determined and measured preoperatively by either spiral or multidetector CT scan
5. ECOG Performance Status ≤1 at study entry
6. Adequate bone marrow haematological function: absolute neutrophil count (ANC) ≥ 1.5 x 109/L AND platelet count ≥ 100 x 109/L AND haemoglobin ≥ 9 g/dL
7. Adequate liver function: total bilirubin ≤ 1.5 x upper limit of normal (ULN) AND aspartate aminotransferase (AST)/alanine aminotransferase (ALT) ≤ 2.5 X ULN
8. Adequate renal function: serum creatinine ≤ 1.5 mg/dL OR creatinine clearance ≥ 60 mL/min in males and ≥50 mL/min in females (calculated according to Cockroft-Gault formula)
9. Serum calcium levels, international normalised ratio (INR) and partial thromboplastin time were within normal limits
10. Female subjects of childbearing potential must have a negative urine pregnancy test result at baseline and practice a reliable method of contraception throughout the study
11. Availability of tumor tissue from basal biopsy for immunoscore and biomarker analysis.
12. Ability to understand study-related patient information and provision of written informed consent for participation in the study

Exclusion Criteria:

1. Evidence of metastatic disease
2. Prior malignancy within the prior 5 years. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer
3. Subjects with active, known or suspected autoimmune disease
4. Subjects with a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of treatment
5. Prior treatment with an anti-PD-1, anti-Programmed Death 1 ligand (PD-L1), anti-PD-L2, or anti-cytotoxic T lymphocyte associated antigen-4 (anti- CTLA-4) antibody
6. Female subjects who are pregnant (positive urine pregnancy test), breastfeeding, or who are of childbearing potential and not practicing a reliable method of birth control
7. Evidence of severe or uncontrolled systemic disease or any concurrent condition which in the investigator's opinion makes it undesirable for the patient to participate in the study, or which would jeopardize compliance with the protocol, or would interfere with the results of the study
8. Patients with a history of cardiovascular or interstitial lung disease and evidence or risk of retinal vein occlusion or central serous retinopathy
9. Inability to regularly access center facilities for logistical or other reasons
10. History of poor co-operation, non-compliance with medical treatment, or unreliability
11. Participation in any interventional drug or medical device study within 30 days prior to treatment start
12. Positive test for hepatitis B virus surface antigen (HBV sAg) or hepatitis C (HCV antibody) with virus ribonucleic acid indicating acute or chronic infection;
13. Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-06-12 (Actual); Primary Completion 2019-06-17 (Actual); Study Completion 2019-09-02 (Actual)

PRIMARY OUTCOMES:
Tolerability and Safety | "up to 5 weeks"
  To determine the feasibility of Nivolumab in the preoperative setting in patients with T3-T4 colon cancer: delay in surgery resection > 21 days after last administration of nivolumab; severe adverse events-NCI CTC-AE Version 4.03 criteria
Clinical Activity | "presurgery"
  Objective Tumor Response Rate (ORR) as defined by Response Evaluation Criteria In Solid Tumors (RECIST)
Predictive Biomarkers | "up to 10 weeks"
  To determine molecular and immunophenotypic changes in tumor and peripheral blood evaluating several biomarkers. Since the identification of new markers for immunotherapy is rapidly evolving, the definitive list of analyses remains to be determined

SECONDARY OUTCOMES:
Pathological Response | "up to 6 weeks"
  To determine the degree of pathologic regression: percentage of patients achieving a pathological complete tumor regression (TRG1)
Clinical efficacy | 3 years
  Relapse-Free Survival
Clinical efficacy | 5 years
  Overall Survival
Toxicities | "up to 3 months"
  Postoperative complications (occurring within 60 days from surgery)
Metabolic Response | "presurgery"
  Metabolic Response by FDG-Positron emission tomography-computed tomography (PET-CT) scan prior to surgery compared to the baseline test.

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Tumori di Napoli - Fondazione G. Pascale, Napoli, Campania, Italy

IPD SHARING:
Plan to Share IPD: No